CLINICAL TRIAL: NCT02150564
Title: Role of 3-D Navigable Ultrasound in Resection of Intra-axial Brain Tumors - A Randomized Controlled Study
Brief Title: 3D Ultra Sound for Resection of Brain Tumors
Acronym: SonoRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Aliasgar V Moiyadi, Prof and Neurosurgeon, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TMC-ACTREC 101
Record Dates: First submitted 2014-05-17; First posted 2014-05-30 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Patients With Resectable Brain Tumors
Keywords: Malignant gliomas; Sono RCT
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Navigation only group (Other): Sonowand system will be used for navigation control arm as well as sononavigation experimental arm.Navigation will be used to plan the craniotomy and throughout the procedure as desired by the operating surgeon. At no point of time however will the Ultrasound be used.
  Interventions: Procedure: Navigation
- SonoRCT Test group (Experimental): Surgery to resect the tumor with the aid of sononavigation. In addition to the navigation function, the Ultrasound will be available at all times. This study will help in assessing the usefulness sononavigation in improving radicality of resection in malignant gliomas and also to access the accuracy of SonoWand in predicting residue.
  Interventions: Device: Sonowand

INTERVENTIONS:
Device: Sonowand — Initially a 2D acquisition will be performed and ultrasound parameters adjusted to obtain the best image resolution. Then anatomical landmarks will be identified if possible and the lesioncharacterized. Once the lesion is identified a rapid 3D-US acquisition will be performed. Tumor resection will proceed guided by the 3D US images using a trackable pointer to navigate. Repeat 3D US images will be obtained as many times as required during the surgery to update the information as tumor debulking proceeds. A final US will be obtained at the end of the procedure and after dural closure
  Arms: SonoRCT Test group
Procedure: Navigation — Routine microneurosurgical procedures would be adopted in all cases.Sonowand system will be used for navigation control arm as well as sononavigation experimental arm. Image registration (on the previously imported DICOM images) will be done on the system and after positioning, patient-toimage registration will be completed. The Registration accuracy will be documented.
  Arms: Navigation only group

SUMMARY:
Phase 3 randomized open labeled trials will evaluate the 3 D navigable ultrasound (SonoWand) in improving the extent of resection in intra-axial brain tumors. All patients will undergo resective surgery. In the experimental arm, a navigable 3 D ultrasound will be used. In the standard arm, only navigation will be used. This study will help in assessing the usefulness sononavigation in improving radicality of resection in malignant gliomas and also to access the accuracy of SonoWand in predicting residue (histopathological correlation).

DETAILED DESCRIPTION:
Routine presurgical evaluation of all patients will be conducted. The preoperative use of steroids, antiepileptics and other medications would be as per standard procedure and would be documented. In addition detailed MRI evaluation will be performed (including contrast enhanced MRI study, diffusion MRI, perfusion MR, MR spectroscopy, dynamic-contrast-enhanced MRI for permeability studies, as well as functional MRI, and tractography if required) not more than 1 week prior to the date of surgery.

Navigation specific MR sequences would be performed in all patients (both arms).

ELIGIBILITY:
Inclusion Criteria:

1. All radiologically-suspected, previously untreated, supratentorial malignant gliomas being considered for debulking surgery.
2. Adults (above 18 years)
3. Eligible for surgical therapy (craniotomy not stereotactic biopsy )
4. Resectability : A lesion would be considered "resectable" if the surgeons feel that all the radiologically imaged lesion can be removed (with reasonable certainty). Only deemed resectable lesions will be included

Exclusion Criteria:

1. Unfit for GA
2. Unwilling for the study
3. Unresectable lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-03; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients where Gross total resection (GTR) achieved | Post operative within 72 hrs.
  Measure: Volumetric MRI - residual tumor (in cc)

SECONDARY OUTCOMES:
Accuracy of US | Post operative within 72 hrours
  Measure: Sensitivity, Specificity, PPV, NPV

OTHER OUTCOMES:
Further resection prompted | Intraoperative
  Whether use of the SonoWand prompted a further resection after the surgeon thought it was complete (Unanticipated residue)
Survival | 3 years
  overall and Progression-free

CONTACTS AND LOCATIONS:
Overall Officials: Aliasgar V Moiyadi, Neurosurgery, Principal Investigator — Prof and Neurosurgeon
Locations (1):
- Advanced Centre for Treatment Research and Education in Cancer, Mumbai, Maharashtra, India